CLINICAL TRIAL: NCT05854381
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Clinical Study to Evaluate the Safety, Reactogenicity and Immunogenicity of the HCMV-HIV Vaccine Candidate VIR-1388 in Adult Participants With Overall Good Health and Without HIV
Brief Title: To Investigate Safety, Reactogenicity and Immunogenicity of VIR-1388 Compared With Placebo in Participants Without HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 142/VIR-1388-V101; 5UM1AI068614-18 (NIH)
Record Dates: First submitted 2023-04-12; First posted 2023-05-11 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: HIV I Infection
Keywords: HIV; Vaccine; CMV; Cytomegalovirus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VIR-1388, 5×10^4 ffu (Experimental): Study intervention will be administered at Day 1 and Day 85 via subcutaneous (SC) injections.
  Interventions: Biological: VIR-1388
- VIR-1388, 5×10^5 ffu (Experimental): Study intervention will be administered at Day 1 and Day 85 via subcutaneous (SC) injections.
  Interventions: Biological: VIR-1388
- VIR-1388, 5×10^6 ffu (Experimental): Study intervention will be administered at Day 1 and Day 85 via subcutaneous (SC) injections.
  Interventions: Biological: VIR-1388
- Placebo (Placebo Comparator): Study intervention will be administered at Day 1 and Day 85 via subcutaneous (SC) injections.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VIR-1388 — VIR-1388 is given by subcutaneous injection
  Arms: VIR-1388, 5×10^4 ffu; VIR-1388, 5×10^5 ffu; VIR-1388, 5×10^6 ffu
Biological: Placebo — The HT Diluent Placebo is HT buffer (20 mM histidine, 10% trehalose-dihydrate, pH 7.2) and contains no active ingredient and will be administered by subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity, and immunogenicity of VIR 1388 in adults in good health without HIV.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled, multicenter study in adults aged 18 to 55 years in overall good health and without HIV. Participants will be enrolled concurrently into 1 of 3 dose levels of VIR-1388 or placebo. The overall study design includes 2 study parts, Part A and Part B. Part A will be a lead-in phase enrolling a limited number of HCMV seropositive persons of non-childbearing potential (PONCBP) with a frequent safety monitoring schedule. Part B will expand enrollment into a broader population of HCMV-seropositive participants, including persons of childbearing potential required to use 2 forms of contraception and maintains a similar overall safety monitoring schedule as Part A . There is an optional long-term follow-up study that would lengthen study participation for up to 3 years post-first dose.

ELIGIBILITY:
Inclusion Criteria:

* In overall good health as determined by medical history, physical exam, and laboratory values
* HIV uninfected
* CMV seropositive
* Willing to use condoms during intercourse for the duration of the study
* Assessed by clinic staff as being low risk for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last protocol visit
* Childbearing status

  * Part A: Only participants of non-childbearing potential
  * Part B: Participants of childbearing potential must be on 2 forms of contraception and not planning on becoming pregnant for the duration of the study

Exclusion Criteria:

* Participant is immunocompromised
* Participant has an autoimmune disorder
* Participants having intimate contact with immunocompromised individuals
* Participants having intimate contact with a pregnant partner or partner planning to become pregnant
* Participants who are breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-11-19 (Actual)

PRIMARY OUTCOMES:
Incidence of unsolicited, treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), new-onset chronic diseases (NOCDs) and medically attended adverse events (MAAEs) | 12 months
  Events will be graded as per the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017
Incidence of solicited local site and systemic reactogenicity events | 14 days after administration of each dose
  Events will be graded as per the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017

SECONDARY OUTCOMES:
Frequency of HIV-1 Mfuse1-specific CD4 T cells | 12 months
  As measured by intracellular cytokine staining (ICS) and flow cytometry
Frequency of HIV-1 Mfuse1-specific CD8 T cells | 12 months
  As measured by intracellular cytokine staining (ICS) and flow cytometry
Memory phenotype of HIV-1 Mfuse1-specific CD4 T cells | 12 months
  As determined by flow cytometry analysis
Memory phenotype of HIV-1 Mfuse1-specific CD8 T cells | 12 months
  As determined by flow cytometry analysis
Number of participants with VIR-1388 vector viremia in plasma | 12 months
  Detected by quantitative polymerase chain reaction(qPCR) of plasma
Number of participants with VIR-1388 vector shedding in saliva and urine | 12 months
  Detected by quantitative polymerase chain reaction(qPCR) of saliva and urine

CONTACTS AND LOCATIONS:
Locations (10):
- United States (6):
  - Alabama CRS, Birmingham, Alabama
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Beth Israel Deconess Medical Center VCRS, Boston, Massachusetts
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CRS, Pittsburgh, Pennsylvania
  - Seattle Vaccine and Prevention CRS, Seattle, Washington
- South Africa (4):
  - Setshaba Research Centre CRS, Soshanguve, Gauteng
  - Perinatal HIV Research Unit, Soweto, Gauteng
  - Isipingo Clinical Research Site, Isipingo, KwaZulu-Natal
  - Chatsworth Clinical Research Site, Overport, KwaZulu-Natal